CLINICAL TRIAL: NCT04631419
Title: Effects of Flapless Laser Corticotomy in Canine Retraction: A Randomized Controlled Trial
Brief Title: Effects of Flapless Laser Corticotomy in Canine Retraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Abubakr Reda Fadeel Ali Bakr, Assistant lecturer , PhD student, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Flapless Laser Corticotomy
Record Dates: First submitted 2020-10-30; First posted 2020-11-17 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Dental Malocclusion; Bimaxillary Protrusion
Keywords: Flapless laser corticotomy; Canine retraction
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Intervention Model Description: The 14 patients maxillary and mandibular arches will be allocated into a split-mouth design, so the sample will be set up each patient to act as his/her own control
Who Masked: Outcomes Assessor
Masking Description: single-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Maxillary flapless laser corticotomy group (Experimental): Flapless laser corticotomy will randomly be assigned to one side of the 14 maxillary arches (experimental side) before canine retraction.
  Interventions: Other: Flapless laser corticotomy; Other: Canine retraction
- Maxillary control group (Active Comparator): Canine retraction will be done on the other side without Laser corticotomy .
  Interventions: Other: Canine retraction
- Mandibular flapless laser corticotomy group (Experimental): Flapless laser corticotomy will randomly be assigned to one side of the 14 mandibular arches (experimental side) before canine retraction.
  Interventions: Other: Flapless laser corticotomy; Other: Canine retraction
- Mandibular control group (Active Comparator): Canine retraction will be done on the other side without Laser corticotomy .
  Interventions: Other: Canine retraction

INTERVENTIONS:
Other: Flapless laser corticotomy — The flapless laser corticotomy will be done by Er, Cr: YSGG laser as a series of circular holes will be made along with the planned position. The depth of laser cutting will be measured and controlled continuously during the operation by the periodontal probe with stopper read to each 3mm depth in addition to a few parts of a millimetre depth into the medullary bone to enhance bleeding. Canine retraction will be started after this procedure.
  Arms: Mandibular flapless laser corticotomy group; Maxillary flapless laser corticotomy group
Other: Canine retraction — canine retraction will be done on 17x25 stst archwire using coil spring adjusted to 150 gm, and miniscrews will be used as an indirect method of anchorage reinforcement

SUMMARY:
This study is conducted to evaluate the effects of flapless laser corticotomy on the rate of canine retraction.

ELIGIBILITY:
Inclusion Criteria:

* Full complement of teeth with no congenitally missing teeth except 3rd molars.
* Minor or no crowding cases requires four premolars extraction, canine retraction & maximum anchorage with bimaxillary dentoalveolar protrusion.
* No history of previous orthodontic treatment
* Clinically healthy patients with no history of drug intake and\or no history for any systemic illness, syndromes, craniofacial deformities.
* Vital teeth with normal periodontium and no root resorption.
* Adequate oral hygiene; probing depth values not exceeding 3 mm across the entire dentition; adequate thickness of the attached gingiva (1-2 mm).
* No radiographic evidence of bone loss.

Exclusion Criteria:

* Systemic disease that might have affected bone formation or density, such as osteoporosis, hyperparathyroidism, or vitamin D deficiency.
* Presence of any local or systemic surgical contraindication.
* Extracted or missing permanent tooth/teeth except for 3rd molars.
* Facial asymmetry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Rate of canine retraction. | 3 months of canine retraction , distance (mm) moved by the canine distally per month
  distal movement of the canine , measurement unit mm divided by time unit month , using scanned digital models

SECONDARY OUTCOMES:
Canine rotation | 3 months, assessed at the beginning of treatment (base line ), and at the end of 3 months of canine retraction
  rotation of canine measured in degrees , after 3 months of canine retraction using scanned digital models
First molar anchorage loss | 3 months, assessed immediately before canine retraction and at the end of 3 months of canine retraction
  mesial movement of first molar measured in mm , after 3 months of canine retraction using scanned digital models
Root resorption | 3 months , assessed at the beginning of treatment (base line ), and at the end of 3 months of canine retraction
  canine root length measured in mm using cone beam CT scans
Periodontal condition | 3 months , immediately before canine retraction , and at the end of 3 months of canine retraction
  assessed using periodontal probe to measure : probing depth in mm
Pulp vitality | 3 months, assessed immediately before canine retraction , and at the end of 3 months of canine retraction
  assessed using thermal (Cold ) test , by application of dry cotton sprayed with ethyl chloride

CONTACTS AND LOCATIONS:
Overall Officials: Abubakr R Bakr, Msc Assistan lecturer, Principal Investigator — Faculty of dentistry , Suez canal university , Ismailia , Egypt
Locations (1):
- Orthodontic department , Faculty of dentistry , Suez Canal University, Ismailia, Egypt

REFERENCES:
- See also: Acceleration of canine movement by laser assisted flapless corticotomy [An innovative approach in clinical orthodontics — http://jbcd.uobaghdad.edu.iq/index.php/jbcd/article/view/530
- See also: Evaluation of piezocision and laser-assisted flapless corticotomy in the acceleration of canine retraction: a randomized controlled trial — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5816528/